CLINICAL TRIAL: NCT02783755
Title: A mHealth Behavioral Cancer Pain Protocol for Medically Underserved Communities.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00065621
Record Dates: First submitted 2016-05-24; First posted 2016-05-26 (Estimated); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: Breast Cancer
Keywords: pain; coping; mhealth; Breast cancer
MeSH Terms: conditions — Breast Neoplasms; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mobile Health Pain Coping Skills Training (mPCST) (Experimental): Mobile Health Pain Coping Skills Training (mPCST) protocol for breast cancer survivors with persistent pain that will produce significant improvements in pain, pain disability, fatigue, physical disability, and adherence to post-treatment lifestyle recommendations that are impacted by pain (i.e., daily activity, self-monitoring of symptoms).
  Interventions: Behavioral: Device: smartphone

INTERVENTIONS:
Behavioral: Device: smartphone — Coping Skills Training for pain will be delivered to participants using video-conferencing

SUMMARY:
The purpose of this study is two-fold. First, the investigator will develop a low-literacy Mobile Pain Coping Skills Training (mPCST) protocol for cancer patients with pain (i.e., therapist manual, patient manual including handouts, and the smartphone materials) as well as a beta version of the basic smartphone components with the assistance of experts in the field. Next, an iterative development design using focus groups with women who have breast cancer and pain accrued from medically underserved areas will be used to refine the developed mPCST protocol and basic smart phone components. The protocol-designed to reduce cancer pain and disability in patients with low literacy in medically underserved areas-will be delivered via tele-video conferencing sessions in the community clinic. The smartphone tools (e.g., simple text messages, images, and preloaded intervention content) will allow the intervention to extend into the patients' homes. The second study purpose is to pilot test the feasibility, acceptability, and efficacy of the developed protocol. The investigator will also obtain an estimate of the effect size of the developed protocol to decrease pain. Focus group data will be managed and evaluated in a systematic format using a grounded theory approach. Data analyses for the pilot testing period of the study will be assessed by examining accrual, attrition, and adherence to the intervention. Simple t-tests will be used to examine pre- to post-intervention differences in pain and the other outcomes of interest. There are minimal risk or safety issues related to this study.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of breast cancer within the last three years
* being >21 years old,
* having a life expectancy of at least 12 months,
* having 1 clinical pain ratings of >3 gathered as part of their routine clinic visits

Exclusion Criteria:

* metastases to the brain,
* presence of a severe psychiatric condition (i.e., psychotic disorder or episode) or a psychiatric condition (e.g., suicidal intent) that would contraindicate safe participation in the study as indicated by the medical chart, treating oncologist, or interactions with the medical/study staff,
* current or past (<6 months) engagement in PCST for cancer.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Change in pain severity will be assessed with the Brief Pain Inventory (BPI). | Baseline and post intervention, approximately 60 minutes
Change in pain Interference will be assessed with the Brief Pain Inventory (BPI) | Baseline and Post Intervention, approximately 60 minutes

SECONDARY OUTCOMES:
Change in self-efficacy for pain control will be assessed with the self-efficacy for pain management subscale of the Chronic Pain Self-Efficacy Scale. | Baseline and Post Intervention, approximately 60 minutes
Change in pain catastrophizing will be assessed with the Coping Strategies Questionnaire. | Baseline and Post Intervention, approximately 60 minutes
Change in Depressive Symptoms:(PROMIS )four-item Depression Scale, a self-report measure of depressive symptoms. | Baseline and Post Intervention, approximately 60 minutes
Change in fatigue | Baseline and Post Intervention, approximately 60 minutes
  The Patient Reported Outcomes Measurement Information System (PROMIS) four-item Fatigue Scale is a self-report measure of fatigue symptoms.
Change in mPCST Acceptability, as measured by participants' engagement | Sessions 2,3,4 and 5
  Patient acceptability of mPCST will be assessed with the Client Satisfaction Questionnaire 10-item version that rates items from 1 = low acceptability and 4 = high acceptability
change in Health-Related Quality of Life | Baseline and Post Intervention, approximately 60 minutes
  The Functional Assessment of Cancer Therapy- General (FACT-G) will be used to assess participants' health-related quality of life. The FACT-G is a 7-item self-report measure that provides participants with a variety of symptoms and concerns.

CONTACTS AND LOCATIONS:
Overall Officials: Tamara J Somers, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No